CLINICAL TRIAL: NCT05638867
Title: A Randomized Controlled Clinical Trial of PARIS Coronary Thrombosis Risk Score Combined With D-dimer to Guide New Oral Anticoagulant Antithrombotic Therapy in Patients With Acute Coronary Syndrome After Percutaneous Coronary Intervention
Brief Title: NOAC Therapy Guided by PARIS Risk Score and D-dimer in Patients With ACS After PCI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Jinqing Yuan, Deputy Director of Coronary Heart Disease Center, Director of Ward 1, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCRC2022003
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Acute Coronary Syndrome
Keywords: Novel Oral Anticoagulant; PARIS risk score; D-dimer; Acute Coronary Syndrome; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Aspirin; Clopidogrel; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Open-label, Two-arm, Randomized Superiority Trial
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study. But while the study is in progress, the grouping information is masked from outcome assessors (CEC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Triple Antithrombotic Therapy: Aspirin (12 months) + Clopidogrel (12 months) + Rivaroxaban (3 months)
  Interventions: Drug: Aspirin + Clopidogrel + Rivaroxaban
- Control Group (Other): Dual Antiplatelet Therapy: Aspirin (12 months) + Clopidogrel (12 months)
  Interventions: Drug: Aspirin + Clopidogrel

INTERVENTIONS:
Drug: Aspirin + Clopidogrel + Rivaroxaban — Triple antithrombotic therapy: aspirin 75-100 mg orally once daily, clopidogrel 75 mg orally once daily, and rivaroxaban 2.5 mg orally twice daily
  Other Names: Triple Antithrombotic Therapy
  Arms: Experimental Group
Drug: Aspirin + Clopidogrel — Dual antithrombotic therapy: aspirin 75-100 mg orally once daily, clopidogrel 75 mg orally once daily
  Other Names: Dual Antiplatelet Therapy
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to compare short-term Triple Antithrombotic Therapy (DAPT + Rivaroxaban) followed by DAPT with standard DAPT in selected ACS patients with high ischemic risk. The main questions it aims to answer are:

* Whether the intervention is effective in reducing ischemic events
* Whether the intervention is safe from increasing bleeding events, especially severe or fatal ones

Participants will be randomized to receive standard DAPT therapy for the entire study duration or low-dose rivaroxaban+DAPT for 3 months, followed by standard DAPT for the rest of the study duration. Patients enrolled should complete 5 follow-ups in the form of clinic visit or telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Acute Coronary Syndrome 1-7 days after initial symptom stabilization,
* Aged 18-65 years old,
* Elevated D-dimer levels (≥0.28 μg/ml) on admission or PARIS coronary thrombosis risk score ≥ 3 points,
* Received Percutaneous Coronary Intervention and not on non-oral anticoagulants,
* Indicated for dual antiplatelet medication

Exclusion Criteria:

* Platelet level below 90 x10^6
* Hemoglobin level is less than 11g/dL
* History of severe bleeding
* History of stroke/TIA
* Severe hepatic/renal insufficiency
* Indicated for anticoagulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3944 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 12 months
  Composite events including all-cause death, myocardial infarction, stroke, ischemia-driven revascularization, stent thrombosis, and systemic embolism

SECONDARY OUTCOMES:
All-cause Death | 12 months
Cardiac Death | 12 months
Myocardial Infarction | 12 months
Stroke | 12 months
Ischemia-driven Revascularization | 12 months
Stent Thrombosis | 12 months
Systemic Embolism | 12 months
Net Adverse Clinical Events | 12 months
  Composite events including MACCE and bleeding

OTHER OUTCOMES:
Bleeding | 12 months
  BARC 3,5 bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Jinqing Yuan, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jia S, Song Y, Yuan D, Wang P, Xu J, Chen Y, Zhang C, Zhao X, Yuan JQ. PARIS coronary thrombosis risk score combined with D-dimer to guide new oral anticoagulant antithrombotic therapy in patients with acute coronary syndrome after percutaneous coronary intervention: study protocol for the PRIDE-ACS trial. BMJ Open. 2025 May 15;15(5):e090126. doi: 10.1136/bmjopen-2024-090126. PMID 40379336